CLINICAL TRIAL: NCT05270044
Title: Adjuvant Encorafenib & Binimetinib vs. Placebo in Fully Resected Stage IIB/C BRAF V600E/K Mutated Melanoma: a Randomized Triple-blind Phase III Study in Collaboration With the EORTC Melanoma Group
Brief Title: Adjuvant Encorafenib and Binimetinib in High-risk Stage II Melanoma With a BRAF Mutation.
Acronym: COLUMBUS-AD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: W00090GE303/EORTC-2139-MG
Record Dates: First submitted 2022-02-14; First posted 2022-03-08 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Melanoma
Keywords: Melanoma; Stage II; BRAFV600E/K; Adjuvant
MeSH Terms: conditions — Melanoma | interventions — encorafenib; binimetinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Encorafenib and Binimetinib
  Interventions: Drug: Encorafenib and Binimetinib
- Arm B (Placebo Comparator): Placebo to match Encorafenib Placebo to match Binimetinib
  Interventions: Drug: Placebo to match Encorafenib ; Placebo to match Binimetinib

INTERVENTIONS:
Drug: Encorafenib and Binimetinib — Encorafenib 450 mg (6 × 75 mg capsules) once daily (QD) and binimetinib 45 mg (3 x 15 mg tablets) twice daily (BID) orally for a maximum of 12 months.
  Other Names: Encorafenib: Braftovi / Binimetinib: Mektovi
  Arms: Arm A
Drug: Placebo to match Encorafenib ; Placebo to match Binimetinib — Encorafenib (6 × 75 mg placebo capsules) QD and binimetinib (3 × 15 mg placebo tablets) BID placebos orally for a maximum of 12 months.
  Arms: Arm B

SUMMARY:
The purpose of the Columbus-AD study is to evaluate the efficacy and safety of 12 months of encorafenib in combination with binimetinib in adjuvant setting of BRAF V600E/K mutant stage IIB/C melanoma versus the current standard of care (surveillance).

DETAILED DESCRIPTION:
This is a randomized triple-blind placebo-controlled international multicenter phase III superiority clinical trial.

Participants with completely resected cutaneous melanoma and documented BRAF V600E/K status by central assay will be randomized 1 to 1 to receive either treatment with encorafenib and binimetinib or their two placebos for 12 months. Patients will be stratified according to the stage of the disease according to AJCC version 8 between:

* stage IIB (i.e., pT3b or pT4a)
* stage IIC (i.e., pT4b).

The long-term evaluation of all endpoints (including information about the occurrence of new treatment-related adverse events, if any) will take place 10 years from the randomization of the last patient.

ELIGIBILITY:
Inclusion Criteria:

Pre-Screening

* Male or female ≥ 18 years of age;
* Surgically resected, with tumour free margins, and histologically/pathologically confirmed new diagnosis of stage II (pT3b-pT4bN0) cutaneous melanomaa;
* Sentinel node (SN) biopsy within 14 weeks from initial diagnosis of melanoma.
* Sentinel node (SN) staged node negative (pN0);
* Available tumour sample for central determination of the BRAF V600E/K mutation.

Screening

* Melanoma confirmed centrally to be BRAF V600E/K mutation-positive;
* Participant still free of disease as evidenced by the required baseline imaging and physical/dermatological assessments performed respectively within 6 weeks and 2 weeks before randomization (Day 1);
* No more than 12 weeks elapsed between full surgical resection (including SLNB) and randomization;
* Recovered from definitive surgery (e.g., complete wound healing, no uncontrolled wound infections or indwelling drains);
* ECOG performance status of 0 or 1;
* Adequate haematological function as defined as Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L and Hemoglobin

  ≥ 9.0 g/dL;
* Adequate renal function as defined as Serum creatinine ≤ 1.5 × ULN; or calculated creatinine clearance ≥ 50 mL/min;
* Adequate electrolytes, defined as serum potassium and magnesium levels within institutional normal limits;
* Adequate hepatic function as defined as Serum total bilirubin ≤ 1.5 x ULN and < 2 mg/dL, Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 2.5 x ULN;
* Adequate cardiac function as defined as LVEF ≥ 50% as determined by MUGA scan or echocardiogram and Mean triplicate QTcF value ≤ 480 msec and no history of QT syndrome;
* Adequate coagulation function, defined as INR ≤1.5× ULN unless the patient is receiving anticoagulant therapy as long as PT or aPTT is within the therapeutic range;
* Negative serum β-HCG test (female patient of childbearing potential only) performed within 3 days prior to Day 1;
* Female patients of child-bearing potential and male patients must agree to follow the protocol's contraception guidance during the treatment period and for ≥30 days after last administration.

Exclusion Criteria:

Pre-screening

* Unknown ulceration status;
* Uveal and mucosal melanoma;
* Clinically apparent metastases (N+/M1);
* Microsatellites, satellites and/or in-transit metastases,
* Local (scar) recurrences.

Screening

* Breast feeding women;
* Pregnant women;
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO;
* History of thromboembolic or cerebrovascular events ≤ 12 weeks prior to randomization;
* History of previous or concurrent malignancy within preceding 3 years or any condition with a life expectancy of less than 5 years;
* Participants with a prior cancer associated with RAS mutation;
* Prior systemic anticancer therapy for melanoma or radiotherapy for melanoma;
* Hypersensitivity to the study drugs or to any of the excipients;
* Participants with severe lactose intolerance (e.g., Rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption);
* Impaired cardiovascular function or clinically significant cardiovascular diseases;
* Neuromuscular disorders that are associated with CK > ULN (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy);
* Non-infectious pneumonitis and Interstitial Lung Disease;
* Positive SARs-CoV-2 or variants of SARs-CoV2 RT-PCR test at screening or suspected to be infected with SARs-CoV2 or variants of SARsCoV2 with confirmation pending;
* Active bacterial, fungal, or viral infection, including, but not limited to HBV, HCV, and known HIV or AIDS-related illness, or an infection requiring systemic therapeutic treatment within 2 weeks prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 815 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2035-05-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | Approximately 4.4 years from the accrual of the first patient.
  RFS is defined as the time between the date of randomization and the date of 1) first recurrence (local, regional, or a distant metastasis), 2) new melanoma that is known to be either ulcerated, thick (Breslow thickness>1 mm) or requiring a treatment other than surgery or 3) death (whatever the cause), whichever occurs first.

SECONDARY OUTCOMES:
Distant metastasis-free survival (DMFS) | Approximately 6.0 years from first patient in
  DMFS is defined as the time between the date of randomization and the date of first distant metastasis or date of death (whatever the cause), whichever occurs first.
Overall survival (OS) | Approximately 10 years from first Patient In.
  OS is defined as time from randomization to the date of death whatever the cause.
Safety - Incidence, nature, severity and seriousness of treatment emergent adverse events (TEAEs) | From the signing of the ICF up to 30 days after end of treatment- approximately 14.5 months
  Incidence nature and severity of adverse events and SAEs graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Safety -Incidence, nature and severity of cutaneous malignancies by dermatological examination | From the signing of ICF to study completion- approximately 10 years from last patient in
  This is to monitor for the possible development of keratoacanthoma and/or squamous cell carcinoma and new primary melanoma, as these have been reported to occur with selective BRAF inhibitor treatment. Incidence, nature and severity of new cutaneous malignancies (kerantoacanthoma, squamous cell carcinoma and new primary melanoma) will be recorded and graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Safety -Incidence of Serious adverse events (SAEs) | From the signing of the ICF to study completion- approximately 10 years from last patient in
  Incidence nature and severity of serious adverse events will be recorded and graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Safety and tolerability - Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes in physical examination | From the signing of the ICF up to 30 days after end of treatment- approximately up to 14.5 months
  Standard physical examinations on cardiovascular, respiratory, gastrointestinal, dermatological, ophthalmological and neurological systems will be performed and will be evaluated based on normal/abnormal and clinical significance observations. Number of participants with TEAEs related to abnormal or clinical significance observations to the physical examinations after the start of study drug will be reported.
Safety and tolerability - Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes in vital signs | From the signing of the ICF up to 30 days after end of treatment- approximately up to 14.5 months
  Clinically notable elevated values: Systolic blood pressure (BP): ≥ 160 mmHg and an increase ≥ 20 mmHg from baseline; Diastolic BP: ≥ 100 mmHg and an increase ≥ 15 mmHg from baseline; Heart rate: ≥ 100 beats/min (bpm) with increase from baseline of ≥ 15 bpm; Body temperature [°C] ≥ 38°C). Clinically notable low values: Systolic BP: <120 mmHg with decrease from baseline of ≥ 20 mmHg; Diastolic BP: < 80 mmHg with decrease from baseline of ≥ 15 mmHg; Heart rate: <50 bpm with decrease from baseline of ≥ 15 bpm; Body temperature [°C]: ≤ 35 °C
Safety and tolerability : Incidence of TEAEs related to notable changes in clinical safety laboratory parameters from baseline. | From the signing of the ICF up to 30 days after end of treatment- approximately up to 14.5 months
  incidence of treatment-emergent adverse events (TEAEs) related to notable changes in clinical safety laboratory parameters from baseline.
  Number of participants with clinically notable shift from baseline in laboratory parameter values based on national cancer institute common terminology criteria (NCI-CTCAE) grade, Version 5.0 will be graded from Grades 1 to 5. Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local or noninvasive intervention indicated. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death. Clinically notable shift is defined as a worsening from baseline by at least 2 grades, or to grade 3 or above.
Safety and tolerability -Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes from baseline of 12-lead electrocardiograms (ECGs) | From the signing of the ICF up to 30 days after end of treatment-approximately up to 14.5 months
  12-lead ECGs will be obtained using an internationally recognized 12-lead cardiograph. Clinically notable ECG values: QT [millisecond (ms)] and QT interval (ms) corrected for heart rate using Fridericia's formula (QTcF) intervals (ms): increase from baseline > 60 ms, new > 450 ms, new > 480 ms, new > 500 ms.
Safety and tolerability - Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes from baseline of echocardiogram or multigated acquisition (ECHO/MUGA) scans. | From the signing of the ICF up to 30 days after end of treatment-approximately up to 14.5 months
  ECHO/MUGA scan assess Left Ventricular Ejection Fraction (LVEF). Changes from baseline of LVEF measurements over time will be reported
Safety and tolerability - Incidence of treatment-emergent adverse events (TEAEs) related to notable or abnormal changes in ophtalmic examination | From the signing of the ICF up to 30 days after end of treatment-approximately up to 14.5 months
  Changes from baseline and worse value on ophthalmic examination over time will be reported.
  a full ophthalmic examination by an ophthalmologist will be performed (at baseline an end of treatment) including best corrected visual acuity (BCVA), slit lamp examination, intraocular pressure (IOP), dilatedfundoscopy and optical coherence tomography (OCT). Retinal examination is required to identify findings associated with retinal pigment epithelial detachments (RPED), serous detachment of the retina and RVO (OCT and angiography).
  the investigator will also monthly monitor visual assesment (general inspection of the eyes, examination of motility and alignment, visual disturbance including diminished central vision, blurred vision or loss of vision).
Safety and tolerability-Treatment emergent adverse events (TEAEs) leading to dose interruption, reduction and discontinuation. | On treatment period - 12 months from randomization.
  Incidence of dose interruptions, dose modifications and discontinuation due to AEs and incidence of AEs requiring additional therapy
Performance status using the Eastern Co-operative Oncology Group (ECOG) performance status scale. | From the signing of the ICF up to 30 days after end of treatment-approximately up to 14.5 months
  Changes from baseline and worse value on Eastern Cooperative Oncology Group (ECOG) Scale with a range from 0 to 5 with lower score mean a lower functional impairment, 5 corresponding to death .
Patient-reported health-related (HRQoL)-European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) . | From the signing of the ICF up to 30 months.
  To determine if there is any change from baseline during the treatment and every 6 months thereafter up to 30 months in the European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) questionnaire scores.
  EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (VAS). The descriptive system has five dimension (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), each is rated according to a five-point verbal rating scale (VRS): 1. no problems, 2. slight problems, 3. moderate problems, 4. severe problems and 5. extreme problems) and translated into a five-digit number that describes the participant's health state
Patient-reported health-related (HRQoL)_European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer Patients (EORTC QLQ-C30) | From the signing of the ICF up to 30 months.
  To determine if there is any change from baseline during the treatment and every 6 months thereafter up to 30 months in the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer Patients (EORTC QLQ-C30) questionnaire scores EORTC QLQ-C30 consists of fifteen multi-item scales: five functional scales (physical, role, cognitive, emotional and social); nine symptom/items scales (fatigue, pain, nausea, vomiting, dyspnea, insomnia, apetite loss, constipation, diarrhae and financial difficulties) and a global health and Quality of Life (QoL) scale. Each scale in the questionnaire will be scored (0 to 100). High scores represents a high health/quality of life
Pharmacokinetic (PK) parameter of encorafenib and its metabolite (LHY746)_Cmin | From randomization up to 11 months
  Minimum serum concentration (Cmin) will be calculated and reported.
Pharmacokinetic (PK) parameter of encorafenib and its metabolite (LHY746)-Cmax | From randomization up to 11 months
  Maximum serum concentration (Cmax) will be calculated and reported.
Pharmacokinetic (PK) parameter of encorafenib and its metabolite (LHY746)_AUC | From randomization up to 11 months
  Area under the curve (AUC) will be calculated and reported.
Pharmacokinetic (PK) parameter of binimetinib and its metabolite (AR00426032)-Cmin | From randomization up to 11 months
  Minimum serum concentration (Cmin) will be calculated and reported
Pharmacokinetic (PK) parameter of binimetinib and its metabolite (AR00426032)-Cmax | From randomization up to 11 months
  Maximum serum concentration (Cmax) will be calculated and reported.
Pharmacokinetic (PK) parameter of binimetinib and its metabolite (AR00426032)-AUC | From randomization up to 11 months
  Area under the curve (AUC) will be calculated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C.J. van AKKOOI, MD, PhD, Study Chair — European Organisation for Research and Treatment of Cancer - EORTC
Locations (155):
- Argentina (8):
  - Centro Oncologico Korben, CABA, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Fundacion CIDEA, Ciudad Autonoma Bs As, Ciudad Autonoma Buenos Aires
  - Sanatorio Britanico S.A., Rosario, Santa Fe Province
  - Instituto de Oncologia de Rosario, Rosario, Santa Fe Province
  - Hospital Aleman, Ciudad Autonoma Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autonoma Buenos Aires
  - Clinica Adventista Belgrano, Ciudad Autonoma Buenos Aires
- Australia (9):
  - Westmead Hospital, Sydney, New South Wales
  - Melanoma Institute Australia, Wollstonecraft, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Adelaide Oncology & Haematolog, Calvary North Adelaide Hospital, North Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Prahran, Victoria
  - Hollywood Private Hospital, Nedlands, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (4):
  - Landeskrankenhaus - Universitaetsklinikum Graz, Graz
  - Krankenhaus der Elisabethinen Linz, Linz
  - Universitätsklinikum St.Pölten-Lilienfeld, Sankt Pölten
  - AKH - Medizinische Universität Wien, Vienna
- Belgium (8):
  - Institut Jules Bordet, Anderlecht
  - ZNA Middelheim, Antwerp
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
  - ZNA, Merksem
  - Vitaz, Sint-Niklaas
  - CHU UCL Namur, Yvoir
- Brazil (10):
  - AMO - Assistência Multidisciplinar em Oncologia, Salvador, Estado de Bahia
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer, Curitiba, Paraná
  - Instituto de Cancer de Londrina, Londrina, Paraná
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - HGB - Hospital Giovanni Battista - Mãe de Deus Center, Porto Alegre, Rio Grande do Sul
  - Instituto de Oncologia Saint Gallen, Santa Cruz do Sul, Rio Grande do Sul
  - CEPON - Centro de Pesquisas Oncológicas de Santa Catarina, Florianópolis, Santa Catarina
  - Fundação Doutor Amaral Carvalho, Jaú, São Paulo
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André, São Paulo
  - A. C. Camargo Cancer Center, São Paulo, São Paulo
- Canada (4):
  - London Health Sciences Centre (LHSC) - Victoria Hospital, London, Ontario
  - Toronto Sunnybrook Hospital, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CIUSSS du Centre Ouest de l'lle de Montreal, Montreal, Quebec
- Czechia (5):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (19):
  - CHU Nice - Hopital de l Archet 2, Nice, Alpes Maritimes
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - CHU de Dijon - Hôpital du Bocage, Dijon, Cote dÝOr
  - CHU de Bordeaux - Hôpital Saint André, Bordeaux, Gironde
  - Institut Claudius Regaud - Oncopole, Toulouse, Haute Garonne
  - Hôpital Ambroise Paré, Boulogne-Billancourt, Hauts De Seine
  - CRLCC Eugene Marquis, Rennes, Ille Et Vilaine
  - CHU Tours - Hôpital Trousseau, Chambray-lès-Tours, Indre Et Loire
  - CHU de Grenoble - Hôpital André Michallon, La Tronche, Isere
  - CHU Nantes - Hôtel Dieu, Nantes, Loire Atlantique
  - Hopital Claude Huriez - CHU Lille, Lille, Nord
  - Hôpital Saint-Louis, Paris, Paris
  - CHU Saint Etienne - Hôpital Nord, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - CAC Clermont-Ferrand Centre Jean Perrin, Clermont-Ferrand, Puy De Dome
  - Centre Hospitalier de Pau - Hôpital François Mitterrand, Pau, Pyrenees Atlantiques
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhone
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen, Seine Maritime
  - Institut Gustave Roussy, Villejuif, Val De Marne
  - CHU Poitiers - Hôpital la Milétrie, Poitiers, Vienne
- Germany (6):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Wuerzburg, Würzburg, Bavaria
  - Elbekliniken Buxtehude GmbH, Buxtehude, Lower Saxony
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Universitaetsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Greece (5):
  - General Hospital of Athens Laiko, Athens
  - Metropolitan Hospital, Neo Faliro
  - Bioclinic Thessaloniki, Thessaloniki
  - Anticancer Hospital of Thessaloniki " Theagenio", Thessaloniki
  - Interbalkan Hospital of Thessaloniki, Thessaloniki
- Hungary (6):
  - Semmelweis Egyetem, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Debreceni Egyetem, Debrecen
  - Petz Aladar Egyetemi Oktato Korhaz, Győr
  - Pecsi Tudomanyegyetem, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Italy (21):
  - IRCCS Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori "Dino Amadori" - IRST, Meldola, Forli - Cesena
  - Ospedale San Vincenzo, Taormina, Messina
  - Istituto Nazionale Tumori Fondazione G. Pascale, Naples, Napoli
  - IRCCS Centro di Riferimento Oncologico, Aviano, Pordenone
  - Istituto Tumori Giovanni Paolo II IRCCS Ospedale Oncologico Bari, Bari
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo
  - Azienda Sanitaria Ospedaliera S.Croce e Carle, Cuneo
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliera di Perugia Ospedale S. Maria della Misericordia, Perugia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Istituto Nazionale Tumori Regina Elena IRCCS, Roma
  - IDI-Istituto Dermopatico dell'Immacolata IRCCS, Roma
  - Policlinico Universitario di Sassari, Sassari
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine
- Netherlands (8):
  - Antoni van Leeuwenhoek, Amsterdam
  - Universitair Medisch Centrum Groningen (UMCG), Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboudumc, Nijmegen
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht
  - Isala, Zwolle
- Norway (2):
  - Ålesund Hospital, Ålesund
  - Oslo University Hospital, Oslo
- Poland (7):
  - Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Gliwice
  - Przychodnia Lekarska Komed, Konin
  - Centrum Onkologii-Instytut im. M. Sklodowskiej-Curie, Krakow
  - Wielkopolskie Centrum Onkologii, Poznan
  - Centrum Medyczne Pratia Poznan, Skórzewo
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
  - Dolnoslaskie Centrum Onkologii, Wroclaw
- Portugal (3):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, EPE, Lisbon
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
- Romania (3):
  - S.C Medisprof S.R.L, Cluj-Napoca
  - S.C Centrul de Oncologie Sf. Nectarie S.R.L, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
- Serbia (6):
  - Clinical Center "Bezanijska kosa", Belgrade
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - Military Medical Academy, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
- South Africa (3):
  - National Hospital Oncology, Bloemfontein, Free State
  - Johese Clinical Research: Midstream, Centurion, Gauteng
  - Sandton Oncology Medical Group, Johannesburg, Gauteng
- Spain (13):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Norrlands Universitetssjukhus, Umeå
- Universitaetsspital Zuerich, Zurich, Switzerland
- United Kingdom (2):
  - Royal Preston Hospital, Preston, Lancashire
  - Northern Centre for Cancer Care, Newcastle upon Tyne, Tyne & Wear

IPD SHARING:
Plan to Share IPD: Yes
Access to de-identified patient-level data in response to scientifically valid research proposals will be provided 30 days after CHMP opinion. All requests from qualified researchers for access to Columbus AD clinical data and information will be managed through a dedicated Pierre Fabre portal.
Supporting Information: Study Protocol, ICF
Time Frame: * Study protocol/Informed Consent Form will be made available in Clinical Trial.gov 30 days after the time of CHMP opinion or up to a maximum of 1 year after the end of the trial whichever is earlier.
  * CSR and SAP: 30 days after the time of CHMP opinion or up to a maximum of 1 year after the end of the trial whichever is earlier.
Access Criteria: Pierre Fabre corporate portal

REFERENCES:
- [Derived] van Akkooi AC, Hauschild A, Long GV, Mandala M, Kicinski M, Govaerts AS, Klauck I, Ouali M, Lorigan PC, Eggermont AM. COLUMBUS-AD: phase III study of adjuvant encorafenib + binimetinib in resected stage IIB/IIC BRAF V600-mutated melanoma. Future Oncol. 2023 Sep;19(30):2017-2027. doi: 10.2217/fon-2023-0414. Epub 2023 Sep 4. PMID 37665297